CLINICAL TRIAL: NCT02652533
Title: Ultrasound Shear Wave Elastography Evaluation of Suspected and Known Biliary Atresia
Status: Completed | Type: Observational
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Siemens Medical Solutions (Industry)
Responsible Party: Sponsor
Other Study IDs: 2015-7320
Record Dates: First submitted 2015-12-18; First posted 2016-01-12 (Estimated); Last update posted 2019-09-23 (Actual); Status verified 2018-03

CONDITIONS: Biliary Atresia
MeSH Terms: conditions — Biliary Atresia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Ultrasound Shear Wave Elastography — The investigators have recently published a very small study in neonates/infants with suspected BA showing that US liver shear wave speed (i.e. - liver stiffness) can differentiate BA from other causes of cholestasis, potentially with a very high degree of accuracy. Additional research is needed to confirm these very preliminary results and determine if liver shear wave speed measurements either before or after (including longitudinally) Kasai can predict key outcomes.

SUMMARY:
The investigators plan to investigate the use of US shear wave elastography (SWE), a newly available imaging technology, in children with suspected/known BA.

DETAILED DESCRIPTION:
The investigators plan a prospective, multi-center study to determine if liver ultrasound shear wave speed measurements acquired at clinical presentation can discriminate biliary atresia (BA) from other causes of liver disease in the setting of neonatal cholestasis. The investigators also plan to determine if liver ultrasound shear wave speed measurements acquired at clinical presentation or longitudinally during the first one-year period after Kasai can predict important long-term outcomes in BA patients.

ELIGIBILITY:
Inclusion Criteria:

* neonatal cholestasis with concern for BA vs. other liver disease direct bilirubin >20% of total or ≥2 mg/dL age <3 months

Exclusion Criteria:

* inability to obtain parent/guardian consent.
* inability to return for follow up visits as required by the study (these patients will be included in aim 1, but will be unable to participate in aim 2).
* no other exclusion criteria.

Max Age: 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: neonatal cholestasis with concern for BA vs. other liver disease direct bilirubin >20% of total or ≥2 mg/dL age <3 months
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2016-09; Primary Completion 2019-01 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
Discrimination of biliary atresia from other liver diseases using ultrasound liver shear wave speed (Aim 1) | 2 years
  The primary outcome measure will be ultrasound shear wave speed of the liver. The investigators will compare the mean liver shear wave speed measurements in children with biliary atresia to other liver diseases. Sensitivity and specificity of ultrasound for diagnosing biliary atresia will be determined using multiple shear wave speed cut-off values.

SECONDARY OUTCOMES:
Predicting long term clinical outcomes in biliary atresia patients using ultrasound liver shear wave speed (aim 2) | 6 years
  Change in shear speed liver over time will be compared between children with biliary atresia versus other liver diseases in order to determine if differences predict important clinical outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Dillman, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (4):
- United States (4):
  - Lucile Packard Children's Hospital/Stanford University, Stanford, California
  - University of Michigan, Ann Arbor, Michigan
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Nationwide Children's, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: No